CLINICAL TRIAL: NCT05400369
Title: A Multicenter, Randomized, Open-Label, Parallel-Controlled Clinical Study to Evaluate the Efficacy and Safety of Sitafloxacin in Adult Subjects With Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Brief Title: A Study to Evaluate the Efficacy and Safety of Sitafloxacin in Adult Subjects With Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSCN-GRV AECOPD-CSIS-001
Record Dates: First submitted 2022-05-27; First posted 2022-06-01 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: COPD Exacerbation Acute
Keywords: Chronic obstructive pulmonary disease; Exacerbation; Sitafloxacin
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — sitafloxacin; Moxifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sitafloxacin (Experimental): Adult participants who will be randomized to receive 100 mg sitafloxacin (2 tablets) orally once a day.
  Interventions: Drug: Sitafloxacin
- Moxifloxacin (Active Comparator): Adult participants who will be randomized to receive 400 mg moxifloxacin (1 tablet) orally every 24 hours.
  Interventions: Drug: Moxifloxacin Hydrochloride

INTERVENTIONS:
Drug: Sitafloxacin — Oral administration, 50 mg tablets
  Other Names: Gracevit
  Arms: Sitafloxacin
Drug: Moxifloxacin Hydrochloride — Oral administration, 400 mg tablets
  Other Names: Avelox
  Arms: Moxifloxacin

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a common, preventable, and treatable disease, that causes obstructed airflow from the lungs that causes persistent obstructive airflow limitation.

Acute exacerbation, especially frequent exacerbation, is associated with an increased risk of death in COPD patients. The most common causes of acute attacks are viral and bacterial infections.

This study will assess the efficacy and safety of sitafloxacin, a quinolone antibacterial drug, in participants with AECOPD.

DETAILED DESCRIPTION:
Clinical evidence suggests that AECOPD may be an important factor in the cause of death in patients with COPD. AECOPD typically presents with increased dyspnea, cough, and sputum volume, or purulent changes in sputum. The most common factors of AECOPD are viral and bacterial infections. Anti-infection agents have shown to be effective in patients with infectious AECOPD.

This study will assess the anti-bacterial drug sitafloxacin in participants with AECOPD. Clinical efficacy is the primary objective of the study. Microbiological validity, symptom relief, magnitude of change in symptom score and inflammatory biomarker, and recurrence rate and safety will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40;
* History of moderate to very severe COPD with a post-bronchodilator Forced Expiratory Volume in One Second/Forced Vital Capacity (FEV1/FVC) < 70% and a post-bronchodilator Forced Expiratory Volume in One Second (FEV1) < 80% of predicted normal value within one year prior to enrollment;
* History of one or more acute exacerbations within one year prior to enrollment;
* At least 6 weeks of stable disease prior to enrollment;
* The acute exacerbation is classified as Anthonisen I (with 3 main symptoms of worsening dyspnea, increased sputum volume and sputum purulence) or II (with sputum purulence and another main symptom);
* Participants can be treated on an outpatient basis after clinical assessment.

Exclusion Criteria:

* Anthonisen III acute exacerbation (Have two major symptoms of worsening dyspnea and increased sputum volume or one of the two major symptoms)
* Hospitalization or intensive care unit (ICU) treatment is required
* Sputum culture within the previous year indicated the presence of pathogenic microorganisms resistant to quinolones
* Quinolone allergy
* History of QTc prolongation, or need for medications to treat QTc prolongation (e.g., Class Ia or Class III antiarrhythmics);
* Definite pulmonary disease other than COPD (asthma, bronchiectasis, active pulmonary tuberculosis, pulmonary embolism, pulmonary fibrosis, lung cancer)
* History of severe cardiovascular disease (e.g., congestive heart failure, clinically significant coronary heart disease, stroke, myocardial infarction and/or stroke within 6 months, clinically significant arrhythmia, previous history of aortic aneurysm or aortic dissection, positive family history, or risk factors (e.g., Marfan syndrome), poorly controlled hypertension (systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg on 2 or more consecutive measurements)
* Severe systemic diseases, such as severe dizziness, headache and other nervous system diseases
* Malignant tumor
* Concomitant or history of tendon disease or myasthenia gravis or Parkinson's disease
* Abnormal liver function, aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) level > 3 times the upper limit of normal, and/or total bilirubin level >2 times the upper limit of normal
* With moderate or severe decline of renal function, endogenous creatinine clearance rate (Ccr) < 50ml/min
* History of seizure, or psychiatric condition that could affect compliance with the protocol, or risk for suicide, or history of alcohol or illicit drug abuse
* Immunocompromised participants using glucocorticoids (total dose equivalent to prednisone 20 mg daily for more than 2 weeks) or immunosuppressive agents or HIV infected participants
* Gastrointestinal disorders that may affect drug absorption (e.g., active Crohn's disease, active ulcerative colitis)
* Pregnant or lactating women or women of childbearing potential who are planning to become pregnant
* Participation in other clinical trials within 3 months prior to screening
* Used antibiotics (including systemic and inhalation) 30 days before enrollment
* Serum potassium < 3.5mmol/L at screening, or repeated hypokalemia that was difficult to correct in the past
* Other reasons that the investigator considered inappropriate to participate in the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
Number of Participants Achieving Clinical Efficacy in Participants With Acute Exacerbation of Chronic Obstructive Pulmonary Disease | End of treatment (approximately Day 10 post-dose)
  Clinical efficacy is divided into clinical cure and clinical ineffective. Clinical cure is defined as the three main symptoms of AECOPD (worsening dyspnea, increased sputum volume and sputum purulence) that disappear or return to the baseline level of stable phase at the end of treatment/discontinuation and no additional systemic antibacterial therapy is required for the target indication.
  Clinical ineffective is defined as the three main symptoms of AECOPD (worsening dyspnea, increased sputum volume and sputum purulence) that persist or incompletely disappear (do not return to the baseline level of stable phase).

SECONDARY OUTCOMES:
Number of Participants Achieving Clinical Efficacy in Participants With Acute Exacerbation of Chronic Obstructive Pulmonary Disease | 1 month post-dose
  Clinical efficacy is divided into clinical cure and clinical ineffective. Clinical cure is defined as the three main symptoms of AECOPD (worsening dyspnea, increased sputum volume and sputum purulence) that disappear or return to the baseline level of stable phase at the end of treatment/discontinuation and no additional systemic antibacterial therapy is required for the target indication.
  Clinical ineffective is defined as the three main symptoms of AECOPD (worsening dyspnea, increased sputum volume and sputum purulence) that persist or incompletely disappear (do not return to the baseline level of stable phase).
Number of Participants Achieving Microbiological Efficacy in Participants With Acute Exacerbation of Chronic Obstructive Pulmonary Disease | End of treatment (approximately Day 10 post-dose)
  Microbiological efficacy is determined by bacterial clearance:
  Clearance is defined as specimens from the original infection site after treatment do not culture pathogenic bacteria from the original infection.
Number of Days With Symptom Relief in Participants With Acute Exacerbation of Chronic Obstructive Pulmonary Disease | From the start of treatment up to relief of three main symptoms of AECOPD (worsening dyspnea, increased sputum volume and sputum purulence), up to 1 month post-dose
  The number of days with symptom relief of the three main symptoms of AECOPD (worsening dyspnea, increased sputum volume and sputum purulence) will be assessed.
Change from Baseline in Each Chronic Obstructive Pulmonary Disease Symptom Score in Participants With Acute Exacerbation of Chronic Obstructive Pulmonary Disease | End of treatment (approximately Day 10 post-dose)
  Chronic obstructive pulmonary disease symptom scores include dyspnea (ranging from 0 [Dyspnea only with strenuous activity] to 4 [Unable to leave home due to severe respiratory distress, or dyspnea when wearing and undressing]), sputum volume (ranging from 0 [no sputum] to 3 [severe]), sputum purulence (ranging from 0 [myxoid sample] to 3 [severe purulent]), cough score (ranging from 0 [no cough] to 3 [severe cough]), fever (ranging from 0 [≤37.0°C] to 3 [>38.0°C], and COPD Assessment Test (CAT) (where questions 1-8, range from a score of 0 [no impact] to 5 [severely impacted]. For all assessments, higher scores indicate worse outcome.
Change from Baseline in Inflammatory Biomarker C-reactive Protein in Participants With Acute Exacerbation of Chronic Obstructive Pulmonary Disease | End of treatment (approximately Day 10 post-dose)
Recurrence Rate of Participants With Acute Exacerbation of Chronic Obstructive Pulmonary Disease | End of treatment (approximately Day 10 post-dose) up to 1 month post-dose
  Recurrence rate is defined as when the clinical outcome of the participant at the end/discontinuation of treatment is determined to be clinically cured, but AECOPD occurs again within 20 days after drug withdrawal due to incomplete anti-infective treatment, the participant develops one or more of the three main symptoms of worsening dyspnea, increased phlegm production, and sputum production, and also has relevant signs of AECOPD, with repeated blood routine, C-reactive protein and other inflammatory indicators, and needs to receive systemic antibacterial drug treatment again, and the pathogenic bacteria belonged to the same strain and serotype as the bacteria originally infected.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director, Study Director — Daiichi Sankyo
Locations (18):
- China (18):
  - Peking University Shougang Hospital, Beijing
  - The Third Xiangya Hospital of Central South University, Changsha
  - The Sixth People's Hospital of Chengdu, Chengdu
  - West China Hospital Sichuan University, Chengdu
  - The First Affiliated Hospital of Dalian Medical University, Dalian
  - Fuyang People's Hospital, Fuyang
  - Nanfang Hospital Southern Medical University, Guangzhou
  - Qilu Hospital of Shandong University, Jinan
  - Gaozhou People's Hospital, Maoming
  - Huadong Hospital Affiliated To Fudan University, Shanghai
  - Shenzhen People's Hospital, Shenzhen
  - Tianjin Medical University General Hospital, Tianjin
  - The Sixth Hospital of Wuhan, Wuhan
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou
  - The First Affiliated Hospital of Hebei North University, Zhangjiakou
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang
  - Henan Provincial People's Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/